CLINICAL TRIAL: NCT02471027
Title: Optimization Research of Early Cervical Caner Treatment
Brief Title: The Clinical Research of Neoadjuvant Chemotherapy Combined Surgery for Locally Advanced Cervical Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Yu mei Wu (Other)
Collaborators: Peking University First Hospital (Other); Peking University Third Hospital (Other); Chinese PLA General Hospital (Other); Beijing Chao Yang Hospital (Other); Beijing Anzhen Hospital (Other); Beijing Shijitan Hospital, Capital Medical University (Other); Peking University People's Hospital (Other)
Responsible Party: Sponsor-Investigator, Yu mei Wu, Beijing Obstetrics and Gynecology Hospital, Capital Medical University, Capital Medical University
Organization: Capital Medical University (Other)
Other Study IDs: D151100001915001
Record Dates: First submitted 2015-05-28; First posted 2015-06-12 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-06

CONDITIONS: Cervical Cancer
Keywords: Locally advanced cervical cancer; Neoadjuvant chemotherapy; Disease-free survival; Overall survival
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Observational Model: Case-Control
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Biospecimen Retention: Samples With DNA — frozen tissue and (or) whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Experimental group: 2009 FIGO staging ⅠB2 or ⅡA2，the treatment is neoadjuvant chemotherapy combined with cervical cancer radical surgery .
  Interventions: Procedure: Neoadjuvant chemotherapy
- control group: 2009 FIGO staging ⅠB2 or ⅡA2，the treatment is cervical cancer radical surgery.

INTERVENTIONS:
Procedure: Neoadjuvant chemotherapy — There is no uniform schemer,commonly used drugs including carboplatin,cisplatin,paclitaxel,vincristine,bleomycin,fluorouracil,ifosfamide,mitomycin,gemcitabine,and so on.Methods including intravenous chemotherapy and artery intervention chemotherapy,also has not been unified.
  Groups: Experimental group

SUMMARY:
This study is a registration study.The main research: the curative effect of neoadjuvant chemotherapy in the treatment of ⅠB2 and ⅡA2 locally advanced cervical cancer.Research group: the neoadjuvant chemotherapy in combination with cervical cancer radical hysterectomy.Control group:cervical cancer radical hysterectomy directly.Main observation indexes is overall survival and disease-free survival.

DETAILED DESCRIPTION:
This study is a multicenter registered study.Selected January 1, 2009 to June 31,2016 ,accepted neoadjuvant chemotherapy combined radical surgery or radical surgery directly as treatment,ⅠB2 and ⅡA2 stage cervical cancer patients at each center to participate in research. Total number of patients is at least 1000 cases.On January 1, 2009 to May 31, 2015 ,collected the baseline data and follow-up information of hospitalized patients ,called a retrospective group.On June 1，2015 to May 31，2016,all the cases into the group take prospective way to collect baseline data (called a prospective group).Mainly collect the follow-up information.

1.The main observation indexes: the overall survival (OS) : the time from treatment for the first time (first day of neoadjuvant chemotherapy or surgery) calculation to the time of death or the time of the last follow-up still alive(about four year).

2.Secondary outcome:

1. 3 year disease-free survival (DFS) : from the operation time or neoadjuvant chemotherapy time calculation for the first time to recurrence/the time or the last follow-up time of death.
2. the quality of life assessment: including EQ-5D health index scale and FSFI scale.
3. the economics indexes: direct and indirect costs.
4. High risk factors of the relapse analysis: lymph node positive rate, cervical local tumor changes after neoadjuvant chemotherapy, pathologic complete response rate after neoadjuvant chemotherapy, tumor pathology classification, tumor stromal infiltration depth, Cut edge positive rate, Vascular infiltration clearance rate, etc.
5. perioperative: operation time, intraoperative blood loss, postoperative complications, postoperative mortality, infections, etc.
6. adverse reactions (prospectie cohort study only) : application WHO anti-cancer drug adverse reaction degree and RTOG/EORTC criteria to evaluate different treatment of adverse reactions.

Subject of supervision organization for clinical research institute is Peking University Clinical Research Institute.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than equal to 18
2. The initial treatment of cervical cancer,the Pathology is squamous cell carcinoma, adenocarcinoma and Adenosquamous carcinoma
3. 2009 FIGO clinical staging IB2, IIA2 stage cervical cancer
4. Patients acceptted the treatment of neoadjuvant chemotherapy combined cervical cancer radical surgery or cervical cancer radical surgery directly
5. Inform consent form

Exclusion Criteria:

1. With severe complications can not tolerate surgery, chemotherapy
2. Patients with distant metastasis
3. With uncontrolled seizures, central nervous system disease or a history of mental disorders, the researchers determine the clinical severity affect clinical research
4. The last five years has a history of other malignant diseases
5. Have received chemotherapy and radiotherapy patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 2009 FIGO clinical staging IB2, IIA2 stage cervical cancer.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-06; Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
overall survival | The average time is up to four year.
  The time from treatment for the first time (first day of neoadjuvant chemotherapy or surgery) calculation to the time of death or the time of the last follow-up(In December 2019) still alive.

SECONDARY OUTCOMES:
3 year disease-free survival (DFS) | The average time is up to three year.
  From the operation time or neoadjuvant chemotherapy time calculation for the first time to recurrence/the time of death or the last follow-up time.

OTHER OUTCOMES:
the quality of life assessment | Before treatment and follow-up period.The average time is up to two year.
  Including EQ-5D health index scale and FSFI scale.
High risk factors of relapse analysis | We get the result after operation.The average time is up to one year.
  The high risk factors of relapse contain:lymgh node positive rate, cervical local tumor changes after neoadjuvant chemotherapy, pathologic complete response rate neoadjuvant chemotherapy, tumor pathology classification, tumor stromal infiltration depth, Cut edge positive rate, Vascular tumor emboli rate, etc.
perioperative indexes | The period of preoperative, intraoperative and postoperative.The average time is up to one year.
  The perioperative indexes contain operation time, intraoperative blood loss, postoperative complications, postoperative mortality, etc.
Adverse reactions | The period of neoadjuvant chemotherapy and postoperative radiotherapy and chemotherapy.The average time is up to one year.
  Application WHO anti-cancer drug adverse reaction degree and RTOG/EORTC criteria to evaluate different treatment of adverse reactions.

CONTACTS AND LOCATIONS:
Overall Officials: Yu M Wu, professor, Principal Investigator — Beijing obstetrics and geynecology hospital
Locations (1):
- Beijing Obstetrics and Gynecology Hospital, Capital Medical University, Beijing, Beijing Municipality, China